CLINICAL TRIAL: NCT03200912
Title: A Multicenter Randomized Doubleblind Vehicle-controlled Parallel Comparison Study to Determine Therapeutic Equivalence of Generic Ingenol Mebutate Gel 0.015% and Picato® Gel 0.015% in Subjects With Actinic Keratosis on the Face or Scalp
Brief Title: An Equivalence Study of Generic Ingenol Mebutate Gel 0.015% and Picato Gel 0.015% in Subjects With Actinic Keratosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 094-8152-301
Record Dates: First submitted 2017-06-14; First posted 2017-06-27 (Actual); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: ACTINIC KERATOSIS
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Picato (Active Comparator): Picato® (ingenol mebutate) gel, 0.15% (Leo Pharma Inc.) [Reference Listed Drug (RLD)]
  Interventions: Drug: Ingenol Mebutate (Picato®)
- Generic Ingenol Mebutate (Experimental): Generic ingenol mebutate gel, 0.15% [Test]
  Interventions: Drug: Generic Ingenol Mebutate
- Vehicle Foam (Placebo Comparator): Vehicle gel of the test product
  Interventions: Drug: Vehicle Foam

INTERVENTIONS:
Drug: Ingenol Mebutate (Picato®) — Brand product
  Other Names: RLD
  Arms: Picato
Drug: Generic Ingenol Mebutate — Generic formulated to have the same therapeutic effect of the brand
  Other Names: Test
  Arms: Generic Ingenol Mebutate
Drug: Vehicle Foam — It does not contain active ingredient. A placebo to test the sensitivity of the active treatments.
  Other Names: Placebo
  Arms: Vehicle Foam

SUMMARY:
The objective of this study was to evaluate the safety and therapeutic equivalence of generic ingenol mebutate gel, 0.015% to Picato gel, 0.015% by establishing the therapeutic comparability of the two active products and the superiority of the two active products over the vehicle gel in the treatment of AK on the face and scalp.

DETAILED DESCRIPTION:
Picato® (ingenol mebutate) gel is the first and only ingenol mebutate product approved by the Food and Drug Administration (FDA) in 2012 for the topical treatment of AKs on the face and scalp (0.015% formulation) and on the trunk and extremities (0.05% formulation). The FDA approved regimen for ingenol mebutate gel, 0.015% for the treatment of AKs on the face and scalp is once-daily application of one unit dose tube for three consecutive days applied to one contiguous skin area of approximately 25 cm2 (e.g., 5 cm x 5 cm).

ELIGIBILITY:
Inclusion Criteria:

* Subject was male or non-pregnant female 18 years of age or older.
* Females must have been post-menopausal, surgically sterile, or using an effective method of birth control. Women of childbearing potential (WOCBP) must have had a negative urine pregnancy test (UPT) at Visit 1/Baseline.
* Subject provided written informed consent.
* Subject had a clinical diagnosis of AK at Visit 1/Baseline with at least four, but no more than eight visible and discrete non-hyperkeratotic, non-hypertrophic AK lesions, each at least 4 mm in diameter, within a contiguous 25 cm2 treatment area ("the Treatment Area") located on the face or scalp.
* Subject was willing and able to apply the test article as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.
* Subject was in good general health and free of any disease state or physical condition that might have impaired evaluation of AK lesions or which, in the investigator's opinion, exposed the subject to an unacceptable risk by study participation.

Exclusion Criteria:

* 1. Subject was pregnant, lactating, or was planning to become pregnant during the study.
* Subject had a location of the selected contiguous 25 cm2 Treatment Area that (a) was within 5 cm of an incompletely healed wound or (b) was in an area containing a lesion that was previously treated with ingenol mebutate.
* Subject had hyperkeratotic, hypertrophic, or large mat-like AKs (e.g., AK >1 cm2 in size) within the contiguous 25 cm2 Treatment Area.
* Subject had more than eight AKs, independent of size, within the selected contiguous 25 cm2 Treatment Area
* Subject had atopic dermatitis, basal cell carcinoma, eczema, psoriasis, rosacea, squamous cell carcinoma, xeroderma pigmentosum, or any other possibly confounding skin conditions within the region of the head that contained the selected Treatment Area (i.e., face or scalp).
* Subject had any skin pathology or condition that, in the investigator's opinion, could have interfered with the evaluation of the test article or required the use of interfering topical, systemic, or surgical therapy.
* Subject was immunosuppressed (e.g., human immunodeficiency virus, systemic malignancy, graft host disease, etc.).
* Subject experienced an unsuccessful outcome from previous ingenol mebutate therapy (an unsuccessful outcome was defined as after a reasonable therapeutic trial with no compliance issues and the topical drug did not work).
* Subject used topical creams, lotions, or gels of any kind within the selected Treatment Area within one day prior to entry into the study.
* Subject had the need or planned to be exposed to artificial tanning devices or excessive sunlight during the study or had used artificial tanners within two weeks of Visit 1/Baseline.
* Subject had used any of the following topical medications on the face or scalp:

  * Corticosteroids within two weeks of Visit 1/Baseline;
  * Keratolytic-containing therapeutic products or medicated or irritant topical salves within two weeks of Visit 1/Baseline, including, but not limited to, alpha hydroxy acids (e.g., glycolic acid, lactic acid etc. >5%), beta hydroxy acid (salicylic acid >2%), and urea >5%;
  * Topical retinoids (e.g., tazarotene, adapalene, tretinoin) within two weeks of Visit 1/Baseline;
  * Light treatments (e.g., psoralen plus ultraviolet A therapy, ultraviolet B) within four weeks of Visit 1/Baseline;
  * Photodynamic therapy within eight weeks of Visit 1/Baseline;
  * 5-fluorouracil, diclofenac, imiquimod, or ingenol mebutate within eight weeks of Visit 1/Baseline; or
  * Other topical therapy for actinic keratosis within 2 cm of the selected contiguous 25 cm2 Treatment Area within eight weeks of Visit 1/Baseline.
* Subject had cryodestruction or chemodestruction, surgical excision, curettage, dermabrasion, chemical peel, or laser resurfacing on the Treatment Area (i.e., face or scalp) within two weeks prior to Visit 1/Baseline.
* Subject used any of the following systemic medications:

  * Corticosteroid therapy within one month;
  * Interferon/interferon inducers, cytotoxic drugs, immuno-modulators, or immunosuppressive therapies within one month;
  * Retinoid therapy within six months prior to Visit 1/Baseline.
* Subject had lesions suspicious for skin cancer (skin cancer not ruled out by biopsy) or untreated skin cancers within the selected contiguous 25 cm2 Treatment Area on the face or scalp.
* Subject was enrolled in an investigational drug or device study.
* Subject used an investigational drug or investigational device treatment within one month prior to Visit 1/Baseline.
* Subject had a history of sensitivity to any of the ingredients in the test articles (see Section 9.4.2).
* Subject had any condition which, in the investigator's opinion, would have made it unsafe or precluded the subject's ability to fully participate in this research study.
* Subject was unable to communicate or cooperate with the investigator due to language problems, poor mental development, impaired cerebral function, or physical limitations.
* Subject was known to be noncompliant or was unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.
* Subject was previously enrolled in the same study.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2016-08-19 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Khatsenko, PhD, Study Director — Actavis Inc.
Locations (23):
- United States (23):
  - Dermatology Specialists, Inc., Oceanside, California
  - Horizons Clinical Research Ctr., LLC, Denver, Colorado
  - The Center for Clinical and Cosmetic Research, Aventura, Florida
  - Moore Clinical Research, Brandon, Florida
  - Savin Medical Group Research Center, Miami Lakes, Florida
  - Tory P. Sullivan, M.D., P.A., North Miami Beach, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Northwest Clinical Trials, Inc., Boise, Idaho
  - Arlington Dermatology, Arlington Heights, Illinois
  - Christie Clinic, LLC, Champaign, Illinois
  - University Dermatology & Vein Clinic, LLC, Darien, Illinois
  - Forefront Dermatology, Carmel, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - The South Bend Clinic,LLC, South Bend, Indiana
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Dermatology Consulting Services, High Point, North Carolina
  - Omega Medical Research, 400 Bald Hill Road, Warwick, RI 02886, Warwick, Rhode Island
  - Palmetto Clinical Trial Services, Fountain Inn, South Carolina
  - Dermatology Associates of Knoxville, PC, Knoxville, Tennessee
  - DermReseach New Braunfels, New Braunfels, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The populations for this study included the Safety Population, the Per-Protocol Population, and the modified Intent-to-Treat (mITT) population.
Groups:
- Generic Ingenol Mebutate: Generic ingenol mebutate gel, 0.015% [Test]
  Generic Ingenol Mebutate: Generic formulated to have the same therapeutic effect of the brand
- Picato (Ingenol Mebutate): Picato® (ingenol mebutate) gel, 0.015% (Leo Pharma Inc.) [Reference Listed Drug (RLD)]
  Ingenol Mebutate (Picato®): Brand product
- Vehicle Gel: Vehicle gel of the test product
  Vehicle Gel: It does not contain active ingredient. A placebo to test the sensitivity of the active treatments.
Period: Overall Study
Arm/Group | Generic Ingenol Mebutate | Picato (Ingenol Mebutate) | Vehicle Gel
Started | 170 | 169 | 168
Completed | 166 | 166 | 164
Not Completed | 4 | 3 | 4
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 4
Not completed — Non-compliance with study drug | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects are from Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Generic Ingenol Mebutate | Picato (Ingenol Mebutate) | Vehicle Gel | Total
Number analyzed (Participants) | 170 | 169 | 168 | 507
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (9.7) | 68.9 (8.6) | 70.2 (9.4) | 69.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 35 | 98
  Male | 139 | 137 | 133 | 409
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 14 | 14 | 43
  Not Hispanic or Latino | 155 | 155 | 154 | 464
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 170 | 168 | 167 | 505
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Complete Clearance of AK Lesions
Description: Treatment success (complete clearance of AK lesions) at Day 57, where complete clearance of AK lesions was defined as having no (zero) clinically visible AK lesions in the Treatment Area
Time Frame: 57 days
Population: AK Complete Clearance Rate at Day 57 (PP population)
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Ingenol Mebutate | Picato (Ingenol Mebutate) | Vehicle Gel
Number analyzed (Participants) | 137 | 144 | 139
Participants | 45 | 44 | 7
Statistical Analysis 1: Comparison: Generic Ingenol Mebutate vs Picato (Ingenol Mebutate); Test type: Equivalence — Primary Efficacy Endpoint - AK Complete Clearance Rates at Day 57 (PP and mITT Populations); Mean Difference (Net) = 2.29, 90% CI 2-sided [-7.55 to 12.14]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of the study start until end of study on Day 57 of the study.
Arm/Group | Generic Ingenol Mebutate | Picato (Ingenol Mebutate) | Vehicle Gel
All-Cause Mortality (participants affected / at risk) | 29/170 | 29/169 | 24/168
Serious Adverse Events (participants affected / at risk) | 2/170 | 0/169 | 2/168
Other Adverse Events (participants affected / at risk) | 29/170 | 29/169 | 24/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Generic Ingenol Mebutate (N=170) | Picato (Ingenol Mebutate) (N=169) | Vehicle Gel (N=168)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation with hospitalization (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Breast cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Ingenol Mebutate (N=170) | Picato (Ingenol Mebutate) (N=169) | Vehicle Gel (N=168)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0
Abdominal pain upper (Eye disorders) | 0 | 1 | 0
Dental caries (Eye disorders) | 0 | 1 | 0
Application site erythema (General disorders) | 1 | 0 | 0
Application site inflammation (General disorders) | 1 | 0 | 0
Application site pain (General disorders) | 6 | 6 | 0
Application site pruritus (General disorders) | 3 | 2 | 0
Application site swelling (General disorders) | 0 | 1 | 0
Breast cellulitis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 3 | 7
Pneumonia (Infections and infestations) | 1 | 0 | 1
Sinusitus (Infections and infestations) | 0 | 3 | 0
Tooth abscess (Infections and infestations) | 1 | 1 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 6
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Headache (Nervous system disorders) | 2 | 1 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Milia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-05-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT03200912/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/12/NCT03200912/SAP_001.pdf